CLINICAL TRIAL: NCT04296682
Title: Impact Of Soft Tissue Manipulation On Dimensional Changes After Posterior Region Extraction: A Randomized Controlled Trial
Brief Title: Impact Of Soft Tissue Manipulation On Dimensional Changes After Posterior Region Extraction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor of Periodontics in Piracicaba Dental School-FOP/UNICAMP, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13838819.1.0000.5418
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Alveolar Ridge Preservation; Connective Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic Extraction Without Gingival Graft (No Intervention): Alveolar closure with elevation of total flaps and simple suture (Silk thread 4.0, Ethicon, Johnson & Johnson, SJC).
- Atraumatic Extraction With Gingival Graft (Experimental): Closure of the alveolus without flap elevation, and placement of a free gingival tissue graft removed from the individual palate.
  Interventions: Procedure: Alveolar Ridge Preservation With Gingival Graft

INTERVENTIONS:
Procedure: Alveolar Ridge Preservation With Gingival Graft — Closure of the alveolus with the placement of a free gingival tissue graft removed from the individual palate.
  Arms: Atraumatic Extraction With Gingival Graft

SUMMARY:
Alveolar preservation seek to avoid multiple surgical interventions to the patient and decrease costs to the patient. In particular, in a Brazilian population where the need for extraction is great, the development of techniques that safely allow a higher quality of rehabilitation is of paramount importance. Thus, this analysis is of great scientific and therapeutic importance. Within the above, the objective is to use an autogenous connective tissue graft in order to eliminate the need to raise the full-thickness flap and compensate for soft tissue deficiencies, which may reduce dimensional losses after extraction, in addition to reducing the cost of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Systemic health (absence of Hypertension and Diabetes);
* Indication of dental extraction of at least 2 teeth (with at least 2/3 of bone support, in the region of premolars or molars with indication for extraction;
* Signature of the consent form;
* Individuals over 18 years old.

Exclusion Criteria:

* Presence of periodontal disease at the time of surgery;
* Pregnant and lactating women;
* Smokers;
* Be under orthodontic treatment;
* Use medication that alters the bone healing process, such as those used to treat osteoporosis and the bisphosphonates group;
* Individuals under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
Minor Alveolar dimensional loss with gingival graft. | 3 months
  Horizontal and vertical bone loss measures after CBCT base and 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, UNICAMP, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No